CLINICAL TRIAL: NCT06357676
Title: Integrated Glofit and Ibrutinib as Novel Immune Therapy Evaluation in Treatment-Naive Mantle Cell Lymphoma (IGNITE MCL): A Phase Ib/II Study of Glofitamab Plus Ibrutinib With Obinutuzumab Pretreatment in MCL Patients ≥ 65 or Ages 18-64 With High-Risk Features
Brief Title: Glofitamab Plus Ibrutinib With Obinutuzumab for the Treatment of Patients With Mantle Cell Lymphoma, IGNITE MCL Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00025355; NCI-2024-01208 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00025355 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2024-04-02; First posted 2024-04-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Specimen Handling; Biopsy; glofitamab; ibrutinib; Magnetic Resonance Spectroscopy; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (glofitamab, ibrutinib, obinutuzumab) (Experimental): Patients receive ibrutinib PO QD on days 1-21 of cycles 1-17. Cycles repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients receive glofitamab IV over 2-4 hours on days 8 and 15 of cycle 2 and then on day 1 of cycles 3-13. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV over 4 hours on cycle 2 day 1 and 2. Additionally, patients undergo echocardiography during screening, bone marrow biopsy on study, and CT scans, FDG PET/CT scans or MRI, and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Echocardiography; Procedure: FDG-Positron Emission Tomography; Biological: Glofitamab; Drug: Ibrutinib; Procedure: Magnetic Resonance Imaging; Biological: Obinutuzumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT scan or FDG PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Procedure: Echocardiography — Undergo echocardiography
  Other Names: EC
Procedure: FDG-Positron Emission Tomography — Undergo FDG PET/CT
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Biological: Glofitamab — Given IV
  Other Names: Anti-CD20 x Anti-CD3 Bispecific Monoclonal Antibody RO7082859; RO 7082859; RO7082859
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759

SUMMARY:
This phase IB/II trial tests the safety, side effects and effectiveness of glofitamab plus ibrutinib with obinutuzumab for the treatment of patients with mantle cell lymphoma (MCL). Glofitamab is in a class of medications called bispecific monoclonal antibodies. It works by killing cancer cells. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). In the body, glofitamab binds to a receptor called CD3 on T-cells (a type of immune cells) and a receptor called CD20 on B-cells, a receptor that is often over-expressed on the surface of cancerous B-cells. When glofitamab binds to CD3 and CD20 receptors, it causes an immune response against the CD20-expressing cancerous B-cells. Ibrutinib is in a class of medications called kinase inhibitors. It works by blocking the action of the abnormal protein that signals cancer cells to multiply. This helps stop the spread of cancer cells. Obinutuzumab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. Glofitamab plus ibrutinib with obinutuzumab may be safe tolerable and/or effective in treating patients with MCL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of treatment with glofitamab and ibrutinib (GLIB) for previously untreated MCL in patients with high risk or age ≥ 65 yrs. (Phase Ib) I. Determine the efficacy of treatment with GLIB for previously untreated MCL in patients with high risk disease or age ≥ 65 yrs. (Phase II)

SECONDARY OBJECTIVES:

I. Assess the overall acute toxicity and tolerability of treatment with GLIB. II. Assess the preliminary efficacy of treatment with GLIB based on clinical response.

III. Assess survival in the absence of progressive disease, recurrence of disease, or death due to any cause after treatment with GLIB.

IV. Assess the duration of clinical response and complete response to treatment with GLIB.

EXPLORATORY OBJECTIVES:

I. Evaluate response to treatment evaluated as minimal residual disease (MRD). II. Evaluate the differential impact of treatment on T cell populations in the tumor microenvironment.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-21 of cycles 1-17. Cycles repeat every 21 days for up to 17 cycles in the absence of disease progression or unacceptable toxicity. Patients receive glofitamab intravenously (IV) over 2-4 hours on days 8 and 15 of cycle 2 and then on day 1 of cycles 3-13. Cycles repeat every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive obinutuzumab IV over 4 hours on cycle 2 day 1 and 2. Additionally, patients undergo echocardiography during screening, bone marrow biopsy on study, and computed tomography (CT) scans, fludeoxyglucose F-18 (FDG) positron emission tomography (PET)/computed tomography (CT) scans or magnetic resonance imaging (MRI), and blood sample collection throughout the study.

After completion of study treatments, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
* Ability to understand the purpose and risks of the study and to provide signed informed consent
* Pathologically confirmed MCL, with documentation of chromosome translocation t(11;14)(q13;q32) and/or overexpression of cyclin D1 in association with other relevant markers (e.g., CD5, CD19, CD20, PAX5). Cyclin D1 negative or t(11,14) negative/SOX 11 positive MCL patients can be enrolled if eligibility criteria are otherwise satisfied
* Age 18-64 with one or more of the following poor risk features defined as:

  * High risk mutational variants including p53 aberrations (mutation[s] by next generation sequencing [NGS] and/or 17p deletion), KMT2D, NSD2, NOTCH1,CDKN2A, NOTCH2, SMARCA4, and CCND1;
  * Blastoid or pleomorphic phenotype;
  * Complex karyotype with ≥ 3 abnormalities (in addition to t(11,14)) on routine karyotyping;
  * Ki67 > 30%;
  * High risk Mantle Cell Lymphoma International Prognostic Index (MIPI) score ≥ 6.2; and/or
  * p53 expression on immunohistochemistry (IHC), defined as ≥ 50%
* Age ≥ 65. For this population, no poor risk features are required to be eligible
* No prior systemic anticancer therapies for MCL
* Presence of radiologically measurable lymphadenopathy and/or extranodal lymphoid malignancy
* Able to provide biosamples for MRD testing and pathology. If fresh tissue is not available, archival samples can be used for some assessments at the discretion of the investigator
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L independent of growth factor support
* Platelets ≥ 100 × 10^9/L (≥ 50 × 10^9/L if bone marrow [BM] involvement), independent of transfusion support in either situation
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 × ULN (unless due to Gilbert's syndrome or of non hepatic origin)
* Estimated creatinine clearance ≥ 50 mL/min by Cockcroft Gault method
* Undetectable hepatitis B virus (HBV) surface antigen (sAg) serology. Confirmed by polymerase chain reaction (PCR) for HBV deoxyribonucleic acid (DNA) if results are disputable
* Undetectable hepatitis C virus (HCV) antigen serology. Confirmed by PCR for HCV ribonucleic acid (RNA) if results are disputable
* Undetectable HIV based on serology. Enrollment will be considered if HIV is controlled with treatment (i.e., undetectable viral load for 6 months prior and the CD4 counts is ≥ 200/µL). Such patients must be willing to modify HIV therapy while on-treatment and during applicable wash-out periods, as needed, to address drug-drug interactions
* Willing and able to participate in all required evaluations and procedures in this protocol including swallowing capsules without difficulty
* Persons of childbearing potential (PCBP): Persons of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [b-hCG]) or urine pregnancy test at Screening and be willing to use approved contraception while on treatment and for the longest following, applicable time period: 18 months after the last dose of obinutuzumab, 2 months after the last dose of glofitamab, 3 months for tocilizumab, or 1 month after the last dose of ibrutinib. Women who are pregnant or breastfeeding are ineligible for this study
* Persons that produce viable sperm: Willingness to use approved contraception while on-treatment and for the longest applicable time period following: 6 months after the last dose of obinutuzumab or 2 months after the last dose of glofitamab, tocilizumab, or ibrutinib
* Willingness to not breastfeed or donate ova or sperm: If obinutuzumab was the last study drug received, the participant must wait for 6 months. Otherwise, patients must agree to wait 3 months for sperm and 1 month for ova donations (and to breastfeed) after the last dose other study drugs
* The effects of GLIB on the developing human fetus are unknown. Should a participant or participant's sexual partner become pregnant or suspect a pregnancy while participating in this study, the individual should inform their treating physician immediately

Exclusion Criteria:

* Previous MCL-directed treatment. Treatment with corticosteroids (up to 20 mg dexamethasone or equivalent daily) is allowed prior to and during the screening period for patients with aggressive clinical behavior. All steroids used for disease control must be discontinued within 7 days before starting study treatment except for doses ≤ 20 mg per day of prednisone or equivalent. Ongoing steroids as premedications or for cytokine release syndrome (CRS) management are allowed on study
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* History of prior malignancy except for the following:

  * Malignancy treated with curative intent and with no evidence of active disease present for more than 2 years before screening and felt to be at low risk for recurrence by treating physician
  * Persons with low grade prostate cancer on a watch and wait strategy are eligible
  * Adequately treated lentigo maligna melanoma without current evidence of disease or adequately controlled nonmelanomatous skin cancer
  * Adequately treated carcinoma in situ without current evidence of disease
  * Ongoing hormonal therapy alone for prior malignancy is allowed
* Concurrent use of cytotoxic chemotherapy; radiotherapy; immunotherapy; hormone therapy (other than contraceptives, hormone-replacement therapy, or megestrol acetate); and biologic agents (other than hematopoietic growth factors, if clinically indicated and used in accordance with manufacture and Investigator recommendations), unless approved by the investigator
* Received systemic immunosuppressive medications (e.g., cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to obinutuzumab infusion with the exception of those described
* Known history of hypersensitivity to

  * Humanized or murine monoclonal antibodies or products
  * A CD3 and / or CD20 antibody
  * Glofitamab
  * Ibrutinib
  * Tocilizumab
* Current or past history of epilepsy, central nervous system (CNS) vasculitis, and neurodegenerative disease
* History of autoimmune disease (e.g., myocarditis, pneumonitis, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Patients with a remote history of, or well controlled, autoimmune disease may be eligible to enroll after consultation with the primary investigator
* History of bleeding risks:

  * Stroke, transient ischaemic attack (TIA),or intracranial hemorrhage within 2 years of first dose of study drug given no remaining neurological deficits
  * Known bleeding diathesis (e.g., hemophilia or von Willebrand disease)
  * Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months prior to cycle 1 day 1 (C1D1)
* Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of first dose of C1D1
* Requires treatment with a strong CYP3A inhibitor/inducer, except for the following:

  * A plan to modify concurrent CYP3A inhibitor/inducer and/or wash-out periods prior to C1D1
  * Topical ketoconazole: Based on its low overall bioavailability, there are no restrictions
* Concurrent participation in another therapeutic clinical trial
* History of confirmed progressive multifocal leukoencephalopathy (PML) or lymphomatous involvement of the CNS
* Known or suspected history of hemophagocytic lymphohistiocystosis (HLH)
* Evidence of ongoing acute or systemic infections (bacterial, fungal, or viral), or any major episode of infection requiring hospitalization or treatment with IV antibiotics (for IV antibiotics this pertains to completion of last course of antibiotic treatment) within 4 weeks of dosing, except localized fungal infections of skin or nails. Subjects may be receiving prophylactic antiviral or antibacterial therapies at the discretion of the investigator
* Receipt of live vaccine within 4 weeks of enrollment or during study treatment period
* Any life-threatening illness, medical condition, or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of ibrutinib capsules, or put the study outcomes at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLT) | At start of cycle 2 day 1 to end of Cycle 3 (each cycle is 21 days)
  The incidence and type of DLT will be reported. Descriptive statistics will be used to report AEs.
Proportion of participants who achieve a complete response (CR) | Start of treatment (Cycle 1 Day 1) to date of first CR, documented at any on-treatment or end-of-treatment (EOT) disease assessment, up to 3 years
  The proportion of patients that achieve a CR will be reported with 95% exact confidence interval (CI). Response to treatment will be evaluated using positron emission tomography/computed tomography (CT) or CT studies and assessed according to Lugano criteria.

SECONDARY OUTCOMES:
Incidence of grade 3 or above adverse events (AEs) | Cycle 1 Day 1 to 30 days after last dose of any study drug
  The incidence of grade 3 or above AEs will be reported with 95% exact CI.
Proportion of patients treated with tocilizumab (TCZ) | Cycle 1 Day 1 to 30 days after last dose of glofitamab (Glt)
  The proportion of patients treated with TCZ will be reported with 95% exact CI.
Number of doses of TCZ per participant | Cycle 1 Day 1 to 30 days after last dose of Glt
  The number of doses of TCZ per participant will be reported with 95% exact CI.
Objective response rate (ORR) | Cycle 1 Day 1 to date of first CR or partial response (PR), documented at any On Treatment or EOT disease assessment, up to 3 years
  ORR (CR + PR) will be defined as the proportion of the efficacy evaluable set that achieves a complete response (CR) or PR at any on-treatment or end of treatment disease assessment. ORR along with 95% CI will be reported.
Progression-free survival (PFS) | Cycle 1 Day 1 to first date of documented progression or death due to any cause, up to 3 years
  PFS will be defined as the time from the first dose of study drug to the first date of documented progression or recurrence or death due to any cause, whichever occurs first. PFS will be summarized descriptively using the Kaplan-Meier method. Median PFS and PFS rates will be estimated with 95% CI if possible.
Duration of response (DOR) | At date of first documented CR/PR to date of progression or death due to any cause, up to 3 years
  DOR will be estimated using the Kaplan-Meier method. Median DOR will be estimated with 95% CI if possible.
Duration of complete response (DOCR) | At date of first documented complete response to first documented progression or death due to any cause, up to 3 years
  DOCR will be estimated using the Kaplan-Meier method. DOCR will be estimated with 95% CI if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States